CLINICAL TRIAL: NCT03889587
Title: Innervation of Vascularized Iliac Transplant Avoids Resorption in Jaw Bone Reconstruction: a Prospective Comparative Clinical Study
Brief Title: Innervation of Vascularized Iliac Transplant Avoids Resorption in Jaw Bone Reconstruction
Acronym: INVITATION
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Collaborators: Örebro University, Sweden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20180506
Record Dates: First submitted 2019-03-11; First posted 2019-03-26 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Bone Resorption; Nerve
Keywords: Jaw reconstruction; Innervation; Bone resorption
MeSH Terms: conditions — Bone Resorption

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Innervation (Experimental): Patients with segmental defects of mandible sized 5 to 12 cm long will be reconstructed using microsurgical iliac or fibula bone flaps. In simultaneous innervated group, neurorrhaphy between the ilioinguinal nerve or fibula flap nerve with inferior alveolar nerve or great auricular nerve will be performed.
  Intervention: Procedure: Innervation
  Interventions: Procedure: Innervation
- Non-innervation (Active Comparator): Patients with segmental defects of mandible sized 5 to 12 cm long will be reconstructed using microsurgical iliac or fibular bone flaps. In traditional noninnervated group, neurorrhaphy will not be performed.
  Intervention: Procedure: Non-innervation
  Interventions: Procedure: Non-innervation

INTERVENTIONS:
Procedure: Innervation — There will be simultaneous innervation of vascularized iliac or fibular bone flaps through neurorrhaphy between the nerves innervating iliac or fibular bones and recipient site.
  Arms: Innervation
Procedure: Non-innervation — This will be the traditional method of vascularized iliac or fibular bone flaps, and neurorrhaphy will not be performed.
  Arms: Non-innervation

SUMMARY:
The purpose of this study is to determine the efficacy of simultaneous innervation to prevent graft bone resorption in maxillofacial reconstruction. It may provide basis for future clinical trials and new strategies for improving the functional reconstruction of large jaw bone defects.

DETAILED DESCRIPTION:
The use of autograft is still the main method for reconstructing large defects of jaw bones. However, the spontaneous resorption of the graft bone is still severe, and hinders the success of dental implant(s) and chewing function even after microsurgical vascularization. But till now, there is no effective prevention method for this major problem. Based on previous studies, the investigators pioneered a simultaneous innervated vascularized iliac bone graft method, through neurorrhaphy between the nerves innervating iliac bone and recipient site. A clinical retrospective study showed that this new method significantly decreases postoperative osteoporosis, and ensures the success of dental implants (Refer to our published article Wang L*, Wei J, Yang X, Yang Z, Sun M, Cheng X, Xu L, Lei D, Zhang C*. Preventing early-stage graft bone resorption by simultaneous innervation: innervated iliac bone flap for mandibular reconstruction. PlastIc Reconstructive Surgery, 2017, 139(5):1152e-1161e, Cover Featured Article).

The investigators intend to randomly divide the vascularized iliac bone graft cases into traditional group without innervation and simultaneous innervation group (through neurorrhaphy between the nerves innervating iliac bone flap and recipient site). The efficacy of simultaneously innervated maxillofacial reconstruction for preventing graft bone resorption will be assessed using bone mineral density test of grafted bone, as a blinded method. The innervation and sensation of the internal oblique abdominis muscle island will be tested using neuroelectrophysiological examination. The recipient nerve having the best effect on preventing bone resorption, will be determined using hierarchical comparison method.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between the age of 17 to 65 years (to avoid possible postmenopause osteoporosis), irrespective of gender.
2. Post resection segmental defect of mandible between 5-9 cm long.
3. Acceptable systemic conditions like nonmenopausal-related osteoporosis, Diabetes mellitus, in controlled normal range.
4. Patients agreeing to sign the informed consent form.

Exclusion Criteria:

1. Advanced malignant tumors.
2. Poor general condition, who can not tolerate vascularized bone flap reconstruction.
3. History of drugs affecting bone metabolism, like bisphosphonates, calcium agents or others.

Ages: 17 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-05-08 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
The efficiency of simultaneously innervated jaw bone reconstruction for preventing graft bone resorption. | Follow-up for 2 years after bone grafting.
  The decreased ratio of the graft bone hounsfield unit calculated by Spiral CT examination ( The hounsfield unit value before bone graft - the hounsfield unit value 1 year after bone graft). It is used to reflect the degree of bone resorption. The efficiency is defined as: the decreased ratio of graft bone hounsfield unit value is less than 10%.
The index of successful innervated reconstruction. | up to 1 year follow-up after bone grafting.
  The innervation and sensation in the muscle island of innervated graft bone flap will be tested using neuroelectrophysiological and needling response examination. The graft bone samples taken by hollow drilling technique during the dental implant(s) procedure will be observed by silver staining. If medullated sensory nerve fibers will be observed, then it indicates successful innervation.

SECONDARY OUTCOMES:
Changes in the outer diameter of the graft bone. | During surgery; After 1 years of bone grafting.
  Measure the outer diameter of the graft bone during the surgery and 1 year after the surgery and compare the difference.

CONTACTS AND LOCATIONS:
Overall Officials: Chenping Zhang, Study Chair — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wang L, Wei JH, Yang X, Yang ZH, Sun MY, Cheng XB, Xu LQ, Lei DL, Zhang CP. Preventing Early-Stage Graft Bone Resorption by Simultaneous Innervation: Innervated Iliac Bone Flap for Mandibular Reconstruction. Plast Reconstr Surg. 2017 May;139(5):1152e-1161e. doi: 10.1097/PRS.0000000000003263. PMID 28445371